CLINICAL TRIAL: NCT04449705
Title: Quality Assessment of a Multifaceted, Perioperative Infection Control Bundle
Status: Withdrawn | Type: Observational
Why Stopped: Hospital didn't use perioperative infection control bundle so study wasn't applicable.
Sponsor: Randy Loftus (Other)
Responsible Party: Sponsor-Investigator, Randy Loftus, Principle Investigator, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202006248
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Perioperative Transmission

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — At the start of each case, the technician will obtain an OR PathTrac kit and will fill out required card indicating the OR number, the surgery date, and the type of surgery. The cards will be placed back into the kit. Sample collection will be directed via use of the kit. The first sample is the adjustable pressure-limiting valve and agent dial of the machine before patient entry (measures terminal cleaning), then provider (attending and assistant) hands after they enter but before patient interaction, then the provider nose and mouth after induction of anesthesia and patient stabilization, then provider hands, then same environmental sites, then provider sites again, then stopcock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical site infections increase patient morbidity and healthcare costs. The Centers for Disease Control and Prevention emphasizes improved basic preventive measures to reduce bacterial transmission and infections for patients undergoing surgery. We conducted a previous study that showed our treatment bundle is highly effective.

Our current study planned to examine patterns/rate of S. aureus transmission to improve feedback widespread implementation of the perioperative infection prevention program at Iowa.

The purpose of this study is to assess the fidelity of the set of interventions in controlling perioperative S. aureus and to provide data feedback via surveillance involving epidemiology of transmission for system optimization.

DETAILED DESCRIPTION:
The operating room schedule will be reviewed each day by the research assistant.

At the start of each case, the technician will obtain an OR PathTrac kit and will fill out required card indicating the OR number, the surgery date, and the type of surgery. The cards will be placed back into the kit. Sample collection will be directed via use of the kit. The first sample is the adjustable pressure-limiting valve and agent dial of the machine before patient entry (measures terminal cleaning), then provider (attending and assistant) hands after they enter but before patient interaction, then the provider nose and mouth after induction of anesthesia and patient stabilization, then provider hands, then same environmental sites, then provider sites again, then stopcock.

A transmission event will be defined as detection of S. aureus pathogens among 2 distinct, epidemiologically-related reservoirs within a surveillance unit. The software platform will process transmission dynamics in order to continually summarize the epidemiology of S. aureus transmission, with results updated daily as case-pair data is continually entered into the program. This information will be continually displayed to identify the most common reservoir of origin, the most common transmission locations (vectors), and involvement of key portals of entry (stopcocks). These will become improvement targets with feedback provided via automated failure mode analysis reports. The research assistant will use the reports to continually optimize the interventions during the observational period.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 years old) patient undergoing surgery requiring anesthesia and placement of a peripheral and/or central intravenous catheter.

Exclusion Criteria:

* <18 years old, Shellfish, iodine, chlorhexidine allergies, no anesthesia and/or placement of peripheral and/or central intravenous catheter required

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery at the University of Iowa
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative transmission of S. aureus | 24 hours
  S. aureus transmission event

CONTACTS AND LOCATIONS:
Overall Officials: Randyt W Loftus, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Request for information must be submitted as a proposal for PI review. Not before 2 years. Use subject to PI review
Supporting Information: Study Protocol
Time Frame: 2 years from study completion
Access Criteria: A written proposal submitted to PI for review